CLINICAL TRIAL: NCT01859858
Title: A Prospective Evaluation of the Effect of Curcumin on Dose-limiting Toxicity and Pharmacokinetics of Irinotecan in Colorectal Cancer Patients
Brief Title: Effect of Curcumin on Dose Limiting Toxicity and Pharmacokinetics of Irinotecan in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LCCC 1227
Record Dates: First submitted 2013-05-17; First posted 2013-05-22 (Estimated); Last update posted 2023-12-04 (Actual); Status verified 2020-06

CONDITIONS: Advanced Colorectal Cancer
Keywords: mCRC (metastatic colorectal cancer); CRC (colorectal cancer); Advanced colorectal cancer; Metastatic colorectal cancer; Colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Curcumin; turmeric extract; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- curcumin + irinotecan (part 1) (Experimental): Oral Curcumin (1, 2, 3,or 4 grams per day) for 4 days prior to irinotecan + 200 mg/m2 irinotecan IV, days 1 and 15
  Interventions: Dietary Supplement: curcumin; Drug: Irinotecan
- curcumin + irinotecan (part 2) (Experimental): MTD oral Curcumin as determined in part 1 + 200 mg/m2 irinotecan IV, days 1 and 15
  Interventions: Dietary Supplement: curcumin; Drug: Irinotecan

INTERVENTIONS:
Dietary Supplement: curcumin
  Other Names: tumeric; Curcuma longa; Meriva
Drug: Irinotecan
  Other Names: Camptosar

SUMMARY:
Curcumin is an extract of the tumeric root that has been shown to have anti-tumor properties in laboratory studies. Curcumin, and its parent spice, turmeric (curcuma longa), are the 4th most commonly purchased dietary supplement in the U.S. Many cancer patients take curcumin during their treatment for cancer because of the purported health benefits.

This research study is designed to learn more about the safety, pharmacokinetics and effectiveness of irinotecan when given in combination with curcumin in patients with metastatic colorectal cancer. The study of how the body absorbs, processes and eliminates drugs is called pharmacokinetics (PK). One of the main purposes of this study is to better understand the interaction between curcumin and irinotecan by measuring levels of irinotecan in the blood (ie. measure irinotecan PK) when a patient also takes curcumin. Information collected from this study could result in improved dosing guidelines and lead to more effective treatment of your cancer with less toxicity.

DETAILED DESCRIPTION:
Treatment Plan

This is a single-center, two-part, open label prospective study to define the maximum tolerated dose (MTD) of curcumin plus irinotecan and the pharmacokinetic effects of curcumin on irinotecan metabolism in patients with advanced colorectal cancer. Each cycle of irinotecan is defined as 28 days, with a dose of irinotecan administered on D1 and D15. The study will have two parts: Part 1 comprises the dose escalation portion of the study and Part 2 comprises the MTD expansion and pharmacokinetic study.

Patients will be recruited from the GI oncology clinic of the North Carolina Cancer Hospital. After obtaining informed consent, patients will be entered into Part 1 of the study until the MTD has been defined. During study Part 1, patients will be given a 4 day run-in of curcumin prior to irinotecan dosing. The planned dose levels of curcumin will be 1, 2, 3, and 4 grams per day. Irinotecan will be dosed at 200 mg/m2 IV on days 1 and 15.46 Additional antineoplastic agents will not be allowed during the trial. Two patients will be enrolled at each dose level until a DLT occurs, beginning with the lowest dose level and increasing the level only after 2 patients have successfully completed a full irinotecan cycle at that dose level.

Part 2 will investigate the effect of curcumin on irinotecan and SN-38 pharmacokinetics. We will expand the cohort of patients at the defined MTD in part 1. Patients will receive irinotecan alone for a single dose (D1). Curcumin, at the MTD, will be started on D11 and continued until the end of the cycle (D28). Irinotecan will be administered again on D15.

Blood samples will be collected on the days of irinotecan infusion (D1 and D15) as follows: prior to treatment with irinotecan (baseline), immediately following the end of irinotecan infusion, and at 0.5, 1, 1.5, 2, 4, 6, and 24 hours following the end of the irinotecan infusion for irinotecan and SN-38 PK.

All patients will continue on curcumin + irinotecan for further cycles until disease progression or toxicity occurs at the discretion of the treating physician (see section 5.6). For patients in study Part 1, we will offer to escalate the curcumin dose to the highest dose level that has been safely completed until an MTD has been estimated.

Treatment Assignment Part 1:

At the end of the screening period, eligible patients are assigned in cohorts of 2 at escalating doses until the first Dose Limiting Toxicity(DLT) is observed. DLT determination will be made based on one cycle in initial cohorts of 2. As much information as possible is used in the initial cohorts of 2. After the first DLT is observed, DLT rates at each dose are estimated using isotonic regression. For that, proportions of DLTs are computed at each dose first, then, if there is a violation of monotonicity, data at the violating dose levels are pooled and new proportions computed. The estimated DLT rate at the current dose is used to determine whether the dose will be increased, decreased or remained unchanged. The dose is to remain unchanged if the estimated DLT rate at the current dose is between [0.17, 0.33]; the dose is decreased if the estimated DLT rate is higher than 0.33; and the dose is increased if the estimated DLT is lower than 0.17. Dose assignment will progress with successful completion of two participants at each dose level until DLT occurs. Dose assignment after the first DLT will be made in collaboration with the study statistician for each patient.

For Part 1, up to 20 patients will be assigned using the algorithm above. The MTD will be estimated when either the highest dose is reached with no DLTs or after 20 patients have completed the algorithm above.

Part 2: After the MTD has been estimated, 10 new patients will be assigned to the "expanded MTD cohort" to estimate PK parameters for irinotecan and SN-38 (active metabolite of irinotecan) with and without curcumin. . The "expanded MTD cohort" might have more than 10 patients if Part 1 sample size is smaller than 20, as long as the total number of patients in the trial does not exceed 30. The estimated MTD might be re-evaluated if the estimated DLT rate at that dose is outside [0.17, 0.33].

ELIGIBILITY:
Inclusion Criteria

1. Age ≥21 years of age (no upper age limit)
2. Histological or cytological documentation of metastatic adenocarcinoma of the colon or rectum. Biopsy of primary tumor alone is adequate if the patient has clear evidence of metastatic disease and/or elevated Carcinoembryonic antigen (CEA) and the treating physician does not feel biopsy of metastatic disease is clinically warranted.
3. Prior therapy with oxaliplatin and a fluoropyrimidine is required. One prior line of therapy with irinotecan is allowed. Prior therapy with an anti-Epidermal Growth Factor Receptor (EGFR) agent is also allowed.
4. Life expectancy of at least 3 months in opinion of treating investigator
5. Eastern Cooperative Oncology Group performance status ≤1 (Appendix B)
6. Adequate bone marrow, renal, and hepatic function, as evidenced by the following within 7 days of treatment initiation with curcumin:

   * absolute neutrophil count (ANC) ≥1,500/mm3
   * platelets ≥100,000/mm3
   * hemoglobin ≥9.0 g/dL
   * serum creatinine ≤1.5 x upper limit of normal (ULN)
   * aspartate aminotransferase (AST) and alanine transaminase (ALT) ≤ 3 x ULN
   * Total bilirubin ≤ 1.5 x ULN
7. Women of childbearing potential and male subjects must agree to use adequate contraception for the duration of study participation. Adequate contraception is defined as any medically recommended method (or combination of methods) as per standard of care.
8. Medical oncologist agrees that four day window on curcumin alone is appropriate/safe prior to start of irinotecan for trial candidate.
9. The subject is capable of understanding and complying with parameters as outlined in the protocol
10. Signed, Institutional Review Board(IRB)-approved written informed consent

Exclusion Criteria:

1. Any prior allergies to curcumin or turmeric.
2. Prior intolerance of irinotecan or necessity for dose reduction greater than 20%
3. Patients who are already known homozygous for the UGT1A1*28 allele (UDP-glucuronosyltransferase 1-1*28), and patients of Asian descent homozygous or heterozygous for the UGT1A1*6 allele will be excluded due to their altered irinotecan metabolism
4. Pregnant or breastfeeding patients. Women of childbearing potential must have a documented negative pregnancy test a maximum of 7 days before start of treatment.
5. History of Gilbert's syndrome
6. Active cardiac disease including any of the following:

   * Congestive heart failure ≥Class 2 according to New York Heart Association [NYHA] (see Appendix C)
   * Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months). Myocardial infarction less than 6 months before start of Day 1 of irinotecan.
   * Cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
7. Ongoing infection > Grade 2 according to NCI Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v. 4.0)
8. Known history of human immunodeficiency virus (HIV) infection
9. Symptomatic metastatic brain or meningeal tumors unless the patient is >3 months from definitive therapy, has a negative imaging study within 4 weeks of irinotecan initiation, and is clinically stable with respect to the tumor at the time of study entry. Also, the patient must not be undergoing acute steroid therapy or taper (chronic steroid therapy is acceptable provided that the dose is stable for one month prior to D1 of treatment under this study)
10. Inability to swallow oral medications or any malabsorption condition
11. Patients with diarrhea CTCAE v4 grade ≥2
12. Unresolved toxicity higher than CTCAE v. 4.0 Grade 1 attributed to any prior therapy/procedure excluding alopecia and oxaliplatin-induced neurotoxicity (which must be ≤ Grade 2)
13. Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
14. Patients unwilling or unable to refrain from use of moderate or strong inhibitors or inducers of Cytochrome P450, family 3, subfamily A (CYP3A) (Appendix A)

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-06; Primary Completion 2016-10-05 (Actual); Study Completion 2016-10-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 28 days
  During Part 1 of study dose escalation will be used to determine the MTD of curcumin based on a DLT rate of 0.25 for the combination with irinotecan.
Pharmacokinetics of irinotecan | 28 days
  The effect of curcumin on irinotecan PK will be evaluated via measurement of plasma Area Under the Curve (AUC) for irinotecan, with and without concomitant curcumin.
Pharmacokinetics of SN-38 | 28 days
  The effect of curcumin on SN-38 PK will be evaluated via measurement of plasma AUC of SN-38, with and without concomitant curcumin.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Asher, MD, MPH, Principal Investigator — University of North Carolina at Chapel Hill Lineberger Comprehensive cancer Center
Locations (2):
- United States (2):
  - IU Simon Cancer Center, Indianapolis, Indiana
  - University of North Carolina at Chapel Hill Lineberger Comprehensive cancer Center, Chapel Hill, North Carolina

REFERENCES:
- See also: UNC Lineberger Website — http://unclineberger.org